CLINICAL TRIAL: NCT05374941
Title: An Interventional Open Feasibility Sleep Study to Determine Effectiveness of StimAire's Injectable and Wearable Neurostimulator in Participants With Obstructive Sleep Apnea
Brief Title: StimAire Sleep Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues related to the intervention
Sponsor: StimAire Australia Pty Ltd (Industry)
Responsible Party: Principal Investigator, Peter Cistulli, Director, Affiliation is Sleep and Breathing Specialist Centre, Sydney, StimAire Australia Pty Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-SA-001
Record Dates: First submitted 2022-03-24; First posted 2022-05-16 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation not synchronized with breathing (Experimental): Participants will be injected with the StimAire Model S Injectable neurostimulator for the hypoglossal nerve, using a wearable without a breathing sensor.
  Interventions: Device: Injectable and wearable neurostimulator for the hypoglossal nerve
- Stimulation during inhalation only (Experimental): Participants will be injected with the StimAire Model S Injectable neurostimulator for the hypoglossal nerve, using a wearable with a breathing sensor.
  Interventions: Device: Injectable and wearable neurostimulator for the hypoglossal nerve

INTERVENTIONS:
Device: Injectable and wearable neurostimulator for the hypoglossal nerve — Temporary placement of injectable and wearable neurostimulator for the hypoglossal nerve

SUMMARY:
The StimAire Model S is intended to treat Obstructive Sleep Apnea (OSA) by stimulating the hypoglossal nerve. The system includes a dedicated neurostimulator and a breathing sensor. The system is to be used in participants diagnosed with moderate to severe Obstructive Sleep Apnea.

The Sponsor will be evaluating the change in Apnea-Hypopnea Index (AHI) when using the StimAire Model S system.

DETAILED DESCRIPTION:
The StimAire Model S is intended to treat Obstructive Sleep Apnea (OSA) by stimulating the hypoglossal nerve. The system includes a dedicated neurostimulator and a breathing sensor. The system is to be used in participants diagnosed with moderate to severe Obstructive Sleep Apnea.

The Sponsor will be evaluating the change in Apnea-Hypopnea Index (AHI) when using the StimAire Model S system.

Single-site controlled AHI measurements both baseline and intervention will be obtained in this open labeled feasibility study. A baseline AHI measurement will be established for each participant, followed by an intervention AHI measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Obstructive Sleep Apnea (defined by AHI > 15 and < 50 per hour of sleep with non-supine AHI>10; with hypopneas defined as greater than 30% reduction in airflow with 3% or greater drop in oxygen saturation). AHI will be determined by full night polysomnography as per guidelines of the American Academy of Sleep Medicine.
2. Age range > 18 years.
3. Difficulty accepting or adhering to, or not desiring of, CPAP therapy.
4. Participant has willingly consented to participate in the study.
5. Participant is willing to remove or have removed facial hair between the base of the neck and the mandible.

Exclusion Criteria:

1. Body mass index > 32 kg/m2. Obese individuals are less responsive to OSA neurostimulation.
2. Documented central or complex sleep apnea > 5 per hour.
3. Participants with pacemaker, defibrillator, or implanted neurostimulators.
4. Hypoxemic and requiring oxygen supplementation.
5. Prior diagnosis of Decompensated cardiac (heart failure [New York heart Association Category III or IV]; or angina) or pulmonary (severe COPD or uncontrolled asthma) disease.
6. Prior diagnosis of any moderate to severe pulmonary artery hypertension.
7. Diagnosis of another sleep disorder in addition to OSA based on PSG (e.g., periodic limb movement arousal index > 10, insomnia, obesity hypoventilation syndrome, or narcolepsy).
8. Hypoglossal nerve palsy on either hypoglossal nerve.
9. Prior diagnosis of neuromuscular disease.
10. Recent or recurring history of recreational drug use leading to tolerance or dependence, at the discretion of the investigators
11. Prior diagnosis of persistent uncontrolled hypertension despite antihypertensive medication use.
12. Any unstable medical or psychiatric comorbidity at the discretion of the investigators
13. Actively taking anticoagulation medication
14. Aspirin taken within 2 weeks prior to injection at the discretion of the investigators
15. Bilateral or unilateral pathology in the submandibular space
16. Actively participating in another clinical trial that to the investigators opinion may compromise this study results.
17. Hypoglossal nerve depth greater than 2.5 cm at the target location of the stimulating electrode as observed on ultrasound display.
18. Tonsil size of 3 or 4 (tonsils visible beyond the pillars or extending to midline) or another anatomical obstruction, at the discretion of the investigators
19. The participant is not appropriate for the regimen for another reason, at the discretion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Change in AHI | Up to 15 Months
  Number of apnea or hypopnea events per hour represented by AHI score

SECONDARY OUTCOMES:
Change in AHI from baseline for stimulation synchronized with inhalation compared to change in AHI for unsynchronized stimulation | Up to 15 Months
  Number of apnea or hypopnea events per hour represented by AHI score

OTHER OUTCOMES:
Percent of successful placements of device | Up to 15 Months
  Number of successful placements of the device

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cistulli, Prof., Principal Investigator — Sleep & Breathing Specialist Centre; Andrew Wignall, Dr., Principal Investigator — Denistone 52 ENT
Locations (1):
- Sleep & Breathing Specialist Centre, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided